CLINICAL TRIAL: NCT02775357
Title: Using the Rakai HIV Risk Index to Measure and Communicate HIV Risk to Create Demand for Safe Male Circumcision: A Randomized Controlled Trial
Brief Title: Measurement of HIV Risk to Create Demand for Safe Male Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rakai Health Sciences Program (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Johns Hopkins Bloomberg School of Public Health (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPP1118591
Record Dates: First submitted 2016-04-07; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: HIV
MeSH Terms: interventions — Weights and Measures; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced HIV counseling and testing (Experimental): In addition to standard HIV testing and counseling,men randomized to this arm received Measurement and communication of HIV risk from the HIV counselors using an index developed and validated through the Rakai community cohort study. Their risk was communicated to them and subsequent HIV risk reduction counseling including male circumcision was given.
  Interventions: Behavioral: Measurement and communication of HIV risk
- Standard HIV testing and counseling (Active Comparator): Men randomized to this arm were given standard HIV testing and counseling following the current Uganda Ministry of Health guidelines. Following the counseling HIV risk reduction counseling including male circumcision was given.
  Interventions: Behavioral: Standard HIV testing and counseling

INTERVENTIONS:
Behavioral: Measurement and communication of HIV risk — Measurement and communication of HIV risk in the context of HIV testing and counseling to inform HIV risk reduction counseling
  Arms: Enhanced HIV counseling and testing
Behavioral: Standard HIV testing and counseling — Participants received HIV testing and counseling following standard Ministry of Health guidelines
  Arms: Standard HIV testing and counseling

SUMMARY:
The study is aimed at testing whether use of a new index to measure risk for HIV in the context of HIV testing and counseling will increase demand for safe male circumcision (SMC) services among HIV-negative non-muslim men in Rakai. We will also study whether use of the index leads to positive sexual behavioral modifications among men. The study will also measure acceptability of the index among men.

DETAILED DESCRIPTION:
Three randomized trials, one of which was conducted in Rakai, Uganda, have shown that safe male circumcision (SMC) reduces HIV acquisition in men by approximately 60%. Recommendations from the World Health Organization (WHO) and the Joint United Nations Programme (UNAIDS) emphasize that SMC should be considered an efficacious intervention for HIV prevention in countries and regions with heterosexual epidemics, high HIV and low male circumcision prevalence.

In Sub Saharan Africa, 14 countries including Uganda have been selected to scale up SMC, for these countries the target is to achieve 80% circumcision prevalence by 2015 and maintain it till 2025. The scale up would avert more than 20 percent of new infections among men and women. However SMC programs are faced with the challenge of low uptake of SMC by older sexually active men who might be at higher risk of HIV. The need to increase SMC coverage among men at high risk of HIV requires tools to measure individual HIV risk.

Rakai Health Sciences Program has received funding to carry out an individual randomized, unblinded, two-arm 1:1 trial comprising a total of 968 men (484 men per study arm) from Rakai Community Cohort Study (RCCS) to assess whether HIV Counseling and Testing (HCT), enhanced with measurement and communication of HIV risk (eHCT), increases uptake of SMC and leads to behavior modification among HIV-negative sexually active men aged 15-49 years in Rakai District, Uganda.

The study is using a risk nomogram developed from the Rakai Community Cohort Study data to measure individual HIV risk in the intervention group and standard HCT in the control arm. All men enrolled will be followed at six months to ascertain circumcision status and collect brief information on sexual behaviors such as number of sex partners, use of alcohol with sex, detailed data on their sexual partners etc.The study will also measure acceptability of the index among men.

ELIGIBILITY:
Inclusion Criteria:

* Uncircumcised, non-muslim, HIV-negative, sexually active in the previous 12 months

Exclusion Criteria:

* Refuses HIV testing, not willing to stay in Rakai for at least 6 months following enrollment or unwilling to be traced

Ages: 15 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 968 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Circumcision status as reported on a questionnaire and confirmed by examination | 6 months
  Circumcision status of men ascertained using a questionnaire and confirmed by examination

SECONDARY OUTCOMES:
Condom use at last non-marital relationship as reported on a questionnaire | 6 months
  Condom use at last non-marital sex ascertained using questionnaire self reports

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kagaayi, Ph.D, Principal Investigator — Rakai Health Sciences Program
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Rakai, Uganda

IPD SHARING:
Plan to Share IPD: No
Data will be published in peer-reviewed journals and at scientific conferences.